CLINICAL TRIAL: NCT06555549
Title: A National, Multicenter, Randomized, Double-blind, Single-dose, Crossover Clinical Trial to Preliminary Evaluate the Efficacy and Safety of DEH113 in the Treatment of Menstrual Cramps Pain Associated With Primary Dysmenorrhea
Brief Title: Efficacy and Safety of DEH113 in the Treatment of Menstrual Cramp Pain in Primary Dysmenorrhea: a Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEH113-P-0123
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEH113 (Experimental): The patient must take two (2) DEH113 tablets in a single dose, if pain.
  Interventions: Drug: DEH113
- Placebo (Placebo Comparator): The patient must take two (2) placebo tablets in a single dose, if pain.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DEH113 — tablets
  Arms: DEH113
Drug: Placebo — tablets
  Arms: Placebo

SUMMARY:
This study aims to evaluate the preliminary efficacy and safety of DEH113 in the Treatment of Menstrual Cramps Pain Associated with Primary Dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent to participate in the study before admission to the study;
* Female patients aged between 16 and 35 years old, inclusive;
* History of regular menstrual cycles, occurring between every 21 to 35 days;
* Clinical history compatible with the diagnosis of primary dysmenorrhea;
* Self-reported history of ≥ 4 painful cycles, with moderate or severe menstrual cramps, in the six (06) months prior to selection for the study.

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea;
* History of non-response to treatment with non-steroidal anti-inflammatory drugs (NSAIDs) to relieve menstrual cramps;
* Onset of primary dysmenorrhea after starting to use oral contraceptives;
* Use of oral contraceptives for < 3 months prior to study selection;
* Use of an intrauterine device (IUD), hormonal implants, or contraceptive injections in the last six (06) months;
* Previous diagnosis or physical examination findings and/or clinical and/or surgical history that may indicate the presence of endometriosis, pelvic inflammatory disease, adenomyosis, mullerian duct malformation, uterine fibroma, cystic ovary and/or pelvic varicocele;
* History of recurrent pelvic and/or lower abdominal pain outside the menstrual period;
* Presence of known allergy or hypersensitivity to the components of the drugs used during the clinical trial;
* History of hypersensitivity reactions, such as asthma attacks or other types of allergic reactions, to acetylsalicylic acid or other NSAIDs;
* Previous diagnosis of glaucoma;
* Previous diagnosis of kidney and/or liver failure;
* Presence of blood dyscrasias and situations of bone marrow suppression;
* Diagnosis of acute intermittent hepatic porphyria;
* Diagnosis of congenital deficiency of glucose-6-phosphate dehydrogenase (G6PD);
* Previous diagnosis of acute intermittent hepatic porphyria;
* Presence of mechanical stenosis in the gastrointestinal tract;
* Previous diagnosis of paralytic ileus or intestinal atony
* Diagnosis of myasthenia gravis;
* Previous diagnosis of severe ulcerative colitis or toxic megacolon complicated with ulcerative colitis
* Treatment with psychoactive drugs (such as for example, antidepressants, antipsychotics, etc.) in the 30 days prior to selection for the study;
* Participants with a history of alcohol or illicit drug use disorder in the last two (02) years;
* Participants with a current medical history of cancer and/or cancer treatment in the last five (05) years;
* Any finding of clinical observation (clinical/physical evaluation) or laboratory condition that is interpreted by the investigating physician as a risk to the participation of the research participant in the clinical trial or the presence of uncontrolled chronic disease(s);
* Participants who are pregnant, nursing, or planning to become pregnant;
* Participation in a clinical research protocol in the last 12 months (CNS Resolution 251, of August 7, 1997, item III, subitem J), unless the investigator judges that there may be a direct benefit to it;

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Sum of Total Pain Relief (TOTPAR) over 0-4, 0-6 and 0-8 hours post-dose | 4, 6 and 8 hours post-dose
  Pain relief will be evaluated considering the Sum of Total Pain Relief (TOTPAR) over 0-4, 0-6 and 0-8 hours post-dose. Pain relief will be evaluate using a Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief).
Sum of Pain Intensity Difference (SPID) over 4, 6 and 8 hours post-dose | 4, 6 and 8 hours post-dose
  Sum of Pain Intensity Difference (SPID) over 4, 6 and 8 hours post-dose. The pain intensity will be assessed using a Categorical 4-point scale (0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain).

SECONDARY OUTCOMES:
Pain intensity (PI) over time | 0, 0.5, 1, 2, 3, 4, 6 and 8 hours post-dose
  PI score assessed 0, 0.5, 1, 2, 3, 4, 6 and 8 hours post-dose
Use of rescue medication | 8 hours post-dose
  Proportion of participants who used rescue medication in the first 8 hours after the first drug intake and time elapsed between the last drug intake and the first administration of rescue medication.
Patients' Global Impression of Change (PGIC) | 8 hours post-dose
  Patients' Global Impression of Change (PGIC) will be assessed after 8 hours post-dose or immediately before the intake of rescue medication

IPD SHARING:
Plan to Share IPD: Undecided